CLINICAL TRIAL: NCT05993884
Title: Phase I Clinical Study on the Safety and Preliminary Efficacy of Allogeneic Endothelial Progenitor Cells (EPCs) Injection in Patients With Acute Ischemic Stroke
Brief Title: Safety and Preliminary Efficacy of Allogeneic Endothelial Progenitor Cells (EPCs) in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: Linfen Central Hospital (Unknown); Peking University Third Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Tiantan Hospital (Other); Linyi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNYX-2020-003
Record Dates: First submitted 2023-04-27; First posted 2023-08-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; EPCs; phase Ⅰ
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental: Cohort 1 (Experimental): 1X level dose of iEPCs
  Interventions: Drug: iEPCs
- Experimental: Cohort 2 (Experimental): 3X level dose of iEPCs or placebo
  Interventions: Drug: iEPCs; Drug: Placebo
- Experimental: Cohort 3 (Experimental): 6X level dose iEPCs or Placebo
  Interventions: Drug: iEPCs; Drug: Placebo
- Experimental: Cohort 4 (Experimental): 10X level dose of iEPCs or placebo
  Interventions: Drug: iEPCs; Drug: Placebo

INTERVENTIONS:
Drug: iEPCs — Patients receive iEPCs IV with the single dose
  Other Names: iPSC EPCs
Drug: Placebo — Patients receive placebo IV with a single dose
  Other Names: iEPCs excipients
  Arms: Experimental: Cohort 2; Experimental: Cohort 3; Experimental: Cohort 4

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-Escalation clinical study to investigate the safety and efficacy of EPCs transplantation in Acute ischemic stroke.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) occurs when blood flow to the brain is blocked by a clot or mechanical event and is the most common type of stroke. However, due to the limitation of time and contraindications, only a few patients with AIS are eligible candidates. Endothelial progenitor cells (EPCs) have the potential to reduce brain damage from AIS. They can effectively repair endothelial cells with vascular injuries by directly differentiating into endothelial cells or releasing corresponding regulatory factors, which is a potentially important means for the prevention and treatment of a series of vascular system disorders. The introduction of induced pluripotent stem cells (iPSCs) technology provides a highly feasible option for clinical application of EPCs. Allogeneic iPSC-EPCs can be produced on a large scale to provide enough cells, fundamentally solving the problem of insufficient dosage, and making them a feasible clinical option for treatment of AIS.

ELIGIBILITY:
Inclusion Criteria:

* 1.Able to provide consent to study or consent is obtained from the patient's legal representative
* 2.Male or females,aged 18 to 80 years
* 3. Subjects with acute ischemic stroke:1) Onset time ≤ 7 days; 2) Imaging confirmed infarction in the blood-supplying area of the internal carotid artery; 3) treated with thrombolysis and/or thrombolysis, or without the above treatment;
* 4.Subjects with NIHSS score between≥6 points and≤24 points at the time of screening
* 5.Eligible patients of childbearing potential(both men and women)if sexually active must agree to use a reliable method of contraception with their partners

Exclusion Criteria:

1. Impaired consciousness (NIHSS score Ia ≥ 2);
2. Disease progression or fluctuation in the subject after the first visit to the screening enrollment, which in the judgment of the investigator has a poor prognosis and will not benefit from this clinical study;
3. Those who have bleeding conversion as assessed by imaging after thrombolysis and/or thrombolysis;
4. History of previous intracranial hemorrhage (within 1 year), arteriovenous malformations, arterial entrapment, aneurysm (≥3 mm in maximum diameter), epilepsy, and history of brain tumor;
5. Abnormalities in major organ function

7. severe respiratory disease that, as assessed by the investigator, may have an impact on the subject's determination of test results (active tuberculosis, chronic obstructive pulmonary disease, interstitial lung disease, severe or critical pneumonia); 8. Uncontrolled hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg) after treatment, which in the judgment of the investigator carries a high risk of bleeding and has a poor prognosis; 9. Those with malignant tumors or a history of malignant tumors; 10. Have an autoimmune disease or are undergoing immunotherapy; 11. Being pregnant or breastfeeding; 12. Allergic to multiple drugs (≥2) or allergic to human albumin; 13. have been alcohol- or drug-dependent in the 6 months prior to the onset of illness or have had an episode of acute alcoholism in the 24 h prior to the onset of illness or have had an episode of Those with acute alcohol intoxication within 24 h; 14. History of psychiatric illness or severe cognitive impairment that may affect the evaluation of neurologic function; 15. Positive for Hepatitis B surface antigen, positive for Hepatitis C virus antibody, positive for syphilis serum antibody or positive for HIV antibody; 16. Being enrolled in a clinical study of another drug; 17. Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the Incidence and severity of adverse events after iEPCs infusion | baseline to 1 year
  Incidence and severity of adverse events assessed by CTCAE V5.0 during the twelve-month study period after iEPCs infusion.

OTHER OUTCOMES:
HLA matching | From enrollment to the end of treatment at 1 year
  the level of HLA matching pairs of donor/recipient
plasma HLA antibody | From enrollment to the end of treatment at 14 days, 1 month and 3 months
  The change from the baseline of plasma HLA antibody will be calculated at Day 14，month 1, month 3 post infusion, as available.
plasma T lymphocytes | From enrollment to the end of treatment at 1 day , 3 days, 7 days, 14 days, 21 days, 1 month , 3 months, 6 months, 9 months, 12 months
  The change from the baseline in plasma T lymphocytes will be calculated at day 1, day 3, day 7, day 14, day 21, month 1, month 3, month 6, month 9, month 12 post infusion, as available.
plasma iEPCs | From enrollment to the end of treatment at 30~40 mins, 1 day, 3 days, 7 days, 14 days, 21 days, 1 month, 2 months, 3 months
  The change from the baseline in plasma iEPCs will be calculated at 30~40 min, day 1, day 3, day 7, day 14, day 21, month 1, month 2, month 3 post infusion, as available.
Modified Rankin Scale, mRS | From enrollment to the end of treatment at 1 month, 3 months, 6 months
  The change from the baseline in mRS will be calculated at month 1, month 3, month 6, as available. The scale is divided into 7 degrees, from 0 (no deficit) to 6 (dead).
National Institute of Health stroke scale, NIHSS | From enrollment to the end of treatment at 1 month, 3 months, 6 months
  The change from the baseline in NIHSS will be calculated at month 1, month 3, month 6 post-treatment, as available. The range of scores is from 0 (normal) to 42.
activity of daily living, ADL | From enrollment to the end of treatment at 1 month, 3 months, 6 months
  The change from the baseline in ADL will be calculated at month 1, month 3, month 6 post-treatment, as available. Every activity will be scored 5 and the range of scores is from 0 (normal) to 5.
cerebral infarct volume | From enrollment to the end of treatment at 7 days and 6 months
  The change from baseline in cerebral infarct volume using MRI will be calculated at day 7, month 6 post-treatment, as available.
vascular endothelial growth factor, VEGF | From enrollment to the end of treatment at 1 day , 3 days, 7 days, 14 days, 21 days, 1 month , 3 months, 6 months, 9 months, 12 months
  Changes of concentration of vascular endothelial growth factor（VEGF）in the serum from the baseline will be calculated at day 1, day 3, day 7, day 14, day 21, month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
brain derived neurotrophic factor，BDNF | From enrollment to the end of treatment at 1 day , 3 days, 7 days, 14 days, 21 days, 1 month , 3 months, 6 months, 9 months, 12 months
  Changes of concentration of brain derived neurotrophic factor (BDNF) in the serum from the baseline will be calculated at day 1, day 3, day 7, day 14, day 21, month 1, month 3, month 6, month 9, month 12 post-treatment, as available.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Allife Medicine （Beijing） Limitied, Beijing, Beijing Municipality
  - Allife, Beijing, Beijing Municipality